CLINICAL TRIAL: NCT03510702
Title: Screening of Epigenetic Biomarkers (miRNA) in the Gingival Sulcus
Brief Title: SCREENING OF EPIGENETIC BIOMARKERS (miRNAs) IN THE GINGIVAL SULCUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, ANA FUENMAYOR GARCÉS, Postgraduate student., University of Valencia
Other Study IDs: H1510580113419
Record Dates: First submitted 2018-04-01; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Periodontal Diseases; Inflammatory Response
Keywords: Epigenetic.; microRNA.; Periodontitis.
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Taking crevicular gingival fluid samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Periodontal patients.: Taking gingival Crevicular fluid.
  Interventions: Diagnostic Test: Levels of epigenetic biomarkers present in the gingival fluid and its possible relationship with bone metabolism.
- Periodontally healthy patients.: Taking gingival Crevicular fluid.
  Interventions: Diagnostic Test: Levels of epigenetic biomarkers present in the gingival fluid and its possible relationship with bone metabolism.

INTERVENTIONS:
Diagnostic Test: Levels of epigenetic biomarkers present in the gingival fluid and its possible relationship with bone metabolism. — Once the anamnesis has been done, all the records corresponding to the Gingival Index and Plaque Index, in both groups are taken.
  Subsequently, samples of gingival crevicular fluid are taken for the screening of epigenetic biomarkers.

SUMMARY:
Epigenetics has produced a high impact in biomedical research and is providing new biomarkers for the diagnosis and prognosis of diseases. In addition, epigenetics is also contributing to analyze the molecular causes underlying diseases, even so periodontal diseases as it has been recently reviewed. In this regard, changes in the methylation of genes codifying for pro-inflammatory and anti-inflammatory cytokines has been previously reported. miRNAs are very promising biomolecules to be used as biomarkers because miRNAs act as signaling molecules and participate in many biological processes, such as cellular development, differentiation, and apoptosis. The high stability of circulating miRNAs in the RNase-rich environment of the bloodstream and also in different biospecimens used in clinical routine, make these biomolecules an optimal source of candidate biomarkers. In fact, miRNAs have demonstrated their value as dynamic biomarkers in a wide variety of human diseases. Therefore, miRNAs can be used for the monitoring of periodontal disease.

The objective of this research is to analyze the levels of bone remodeling RANKL / OPG biomolecular markers, and the epigenetic regulation of these proteins to identify promising biomarkers of periodontal disease.

Material and Methods. Levels of RANKL and OPG will be measured in the gingival crevicular fluid (GCF) to assess the state of bone. These samples will be sent to the lab for quantification by ELISA method.

Furthermore, new epigenetic biomarkers based on the identification of high stable microRNAs will be identified by qRT-PCR in GCF as feasible tools for diagnosis and monitoring of wide range of disease, including periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

Group of periodontal patients:

1. Clinical criteria: at least 3 locations in unirradicular teeth with PD 6 mm. 3 samples will be taken from each of these 3 locations (9 total samples). Third molars are not included in the study.
2. Patients not treated periodontally.
3. 30-60 years.

Periodontally healthy group:

1. Absence of clinical and radiographical periodontal pathology.

Exclusion Criteria:

* Group of periodontal patients:

  1. Aggressive Periodontal Disease (Armitage, 1999).
  2. Patients with controlled periodontal disease with plaque and gingival indexes ≤20%.
  3. Patients with systemic diseases or taking medications that alter bone metabolism (Osteoporosis, arthritis, hormonal treatment, bisphosphonates, anti-inflammatory, immunosuppressants, etc ...).
  4. Patients with antibiotic, anti-inflammatory or contraceptive treatment in the previous 3 months or taking antiaggregants in the last 7 days before taking the sample.
  5. Smokers (> 10 cig. /day).
  6. Pregnant or breast-feeding.

Periodontally healthy group:

1. Patients with systemic diseases or taking medications that alter bone metabolism (Osteoporosis, arthritis, hormonal treatment, bisphosphonates, anti-inflammatory, immunosuppressant...).
2. Patients with antibiotic, anti-inflammatory or contraceptive treatment in the previous 3 months or taking antiaggregants in the last 7 days before taking the sample.
3. Smokers (> 10 cig/day).
4. Pregnant or breast-feeding.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients attending to the university who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
microRNA in gingival crevicular fluid (physiological parameter). | 2 years.
  Insert the Perio Paper® tip in gingival sulcus until resistance is felt and leave it for 30 seconds.

SECONDARY OUTCOMES:
Probing depth. | 2 years.
  Probing depth will be measured in six sites (disto-buccal, mid-buccal, mesio-buccal, disto-palatal, mid-palatal and mesio- palatal) of every teeth with a Williams Probe PQ-OW 208 396. This probe is used by gently hanging pressure into a pocket measuring 20 grams in weight.
Bleeding on probing. | 2 years.
  Full mouth bleeding score (FMBS) will be calculated based on scores of 0 (no bleeding) or 1 (bleeding) after probing for PD. The usual thing to do is to measure at 4 points for each tooth but we have modified the index and we valorate them at 6 points. (disto-buccal, mid-buccal, mesio-buccal, disto-palatal, mid-palatal and mesio- palatal).
Clinical recession. | 2 years.
  Clinical recession will be measured in the same six sites as before between the Amelocemental junction and the gingival margin.
Plaque score of Silness y löe: (1964) | 2 years.
  The Plaque will be scored as follows:
  Score 0 = No plaque
  Score 1 = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  Score 2 = Moderate accumulation of soft deposits within the gingival pocket, or on the tooth and gingival margin, which can be seen with the naked eye.
  Score 3 = Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  The usual thing to do is to evaluate at 4 points for each tooth but we have modified the index and we will evaluate at 6 points. (disto-buccal, mid-buccal, mesio-buccal, disto-palatal, mid-palatal and mesio- palatal)
Dental movility of Mïller 1950 | 2 years.
  Class I
  Up to 1 mm of movement in a horizontal direction.
  Class II Greater than 1 mm of movement in a horizontal direction. Class III
  Excessive horizontal movement and vertical movement.
Furcation affection. | 2 years.
  Class I:
  The level of bone loss allows for the insertion of the periodontal Nabers probe into the concavity of the root trunk. Furcation defect is less than 3 mm is depth.
  Class II The level of bone loss allows for the insertion of a periodontal probe into the furcation area between the roots. Furcation defect is at least 3 mm in depth (and thus, in general, surpassing half of the buccolingual thickness of the tooth) but not through-and-through (i.e. there is still some interradicular bone attached to the angle of the furcation.
  15
  Class III The level of bone loss allows for "through and through" access of the furcation area. Buccal to lingual on lower molars. Buccal to mesio-palatal and disto-palatal on upper molars. Furcation defect encompassing the entire width of the tooth so that no bone is attached to the angle of the furcation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Fuenmayor Garcés, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided